CLINICAL TRIAL: NCT02179411
Title: Study of the Renal Perfusion in Healthy Volunteers and Renal Transplant Recipients During an Orthostatic Stress
Acronym: ortho_rein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-P2009-01
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2009-04

CONDITIONS: Safe Volunteers; Kidney Transplant Recipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- healthy volunteers (Active Comparator): healthy volunteers
  Interventions: Other: tilt test
- renal transplant recipients (Active Comparator): renal transplant recipients
  Interventions: Other: tilt test
- renal transplant recipients grave (Active Comparator): renal transplant recipients grave
  Interventions: Other: tilt test

INTERVENTIONS:
Other: tilt test

SUMMARY:
Autonomic nervous system contributes to the regulation of renal blood flow, affected by upright posture. Kidney transplantation implies sympathetic denervation. The aim of this study is to compare the renal vascular response in volunteers and renal graft recipients to an orthostatic stress induced by a head-up tilt test. Renal peripheral resistances are assessed by echo Doppler. The sympathetic nervous system activity is evaluated by plasma concentrations of catecholamine before and after the head-up tilt test.

ELIGIBILITY:
Inclusion Criteria:

- Healthy volunteers Male or female, within 18 and 50 year old Caucasian type

No cardiovascular risk factor:

Body mass index below 25 kg/m2 No smoking No dyslipidemia No diabetes No kidney disease or chronic renal failure No medication Electrocardiogram: normal Arterial blood pressure: normal Plasma creatinine clearance equivalent to 50mL/min or more (Cockroft formula) No proteinuria and no hematuria Able to understand the purpose of the study and sign the informed consent

- Renal graft recipients Male or female, within 18 and 50 year old Caucasian type About a year after the first renal allograft Body mass index below 25 kg/m2 No smoking No dylipidemia No diabetes Arterial blood pressure controlled Electrocardiogram: normal Plasma creatinine clearance equivalent to 50mL/min or more (Cockroft formula) Able to understand the purpose of the study and sign the informed consent

Exclusion Criteria:

* Healthy volunteers Creatinine clearance < 50 mL/min (Cockroft formula) More than 2 syncopes a year Pregnancy
* Renal graft recipients Creatinine clearance < 50 mL/min (Cockroft formula) Second renal allograft or more More than 3 antihypertensive treatments Beta adrenoreceptors blockers Acute rejection More than 2 syncopes a year

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of vascular resistance standing in renal transplant subjects compared with healthy subjects. | three years
  Evaluation of vascular resistance standing in renal transplant subjects compared with healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU d'Angers, Angers, France